CLINICAL TRIAL: NCT06363604
Title: Randomized Controlled Study of Atrial Posterior Wall Isolation (PWI) Assisted by Vein of Marshall Ethanol Infusion (VOMEI) and Pulmonary Vein Isolation in Persistent Atrial Fibrillation Ablation
Brief Title: Evaluation of PWI Assisted by Marshall Ethanolization in Ablation of Persistent Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHEC-C-2023-128-2
Record Dates: First submitted 2024-01-21; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A total of 260 participants with persistent AF who undergo radiofrequency catheter ablation and received VOMEI + PVI will be randomized assigned to two groups at 1:1 ratio.
  Group 0 (Control): VOMEI + PVI + linear ablation of mitral isthmus. Group 1 (Experimental): VOMEI + PVI + linear ablation of mitral isthmus + PWI
Who Masked: Participant
Masking Description: This study used a single-blind design for the subjects. A statistician created a random sequence of numbers using a randomization scheme. The sequence was then placed in opaque coded envelopes and sealed in numerical order. When a patient met the inclusion and exclusion criteria and was assigned a number, the researcher notified the manager to obtain the corresponding envelope and perform the intervention according to the grouping plan inside the envelope. Group 0 correspond to the control group not receiving PWI isolation, while group 1 correspond to the experimental group for PWI isolation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOMEI + PVI + linear ablation of mitral isthmus + PWI (Experimental): Acquisition of left atrial posterior wall isolation by linear ablation of LA roof and bottom line, in addition to routine strategy with vein of Marshall ethanol infusion, isolation of bilateral pulmonary veins and linear ablation of mitral isthmus.
  Interventions: Procedure: VOMEI + PVI + linear ablation of mitral isthmus; Procedure: Posterior wall isolation
- VOMEI + PVI + linear ablation of mitral isthmus (Active Comparator): Routine strategy with vein of Marshall ethanol infusion, isolation of bilateral pulmonary veins and linear ablation of mitral isthmus. Left atrial posterior wall not isolated.
  Interventions: Procedure: VOMEI + PVI + linear ablation of mitral isthmus

INTERVENTIONS:
Procedure: VOMEI + PVI + linear ablation of mitral isthmus — The CS angiography is firstly performed to visualize the vein of Marshall. The ethanol infusion by anhydrous alcohol is then performed by using a guidewire and an OTW ballon. For radiofrequency catheter ablation, the standard procedure of pulmonary vein isolation is performed. All the enrolled persistent AF patients perform the routine linear ablation of mitral isthmus.
Procedure: Posterior wall isolation — PWI is additionally performed for experimental group with linear ablation of LA roof and bottom line, and verified by mapping with a multielectrode catheter.
  Other Names: PWI
  Arms: VOMEI + PVI + linear ablation of mitral isthmus + PWI

SUMMARY:
This is a prospective, randomized controlled, single-blind, multi-center clinical trial study aiming to investigate whether the strategy of posterior wall isolation (PWI) assisted by vein of Marshall ethanol infusion (VOMEI) could improve the success rate of persistent atrial fibrillation ablation.

DETAILED DESCRIPTION:
A total of 260 participants with persistent AF who undergo radiofrequency catheter ablation and received VOMEI + PVI will be randomized assigned to two groups at 1:1 ratio.

Group 1: VOMEI + PVI + linear ablation + PWI; Group 2: VOMEI + PVI +linear ablation. The major endpoint (efficacy endpoint) is the recurrence of atrial tachyarrhythmias between 3-12 months during follow-up. The secondary endpoint (safety endpoint) is the occurrence of procedural complications.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-85 years old;
2. Symptomatic, non-valvular persistent atrial fibrillation (atrial fibrillation duration ≥1 week), and refractory to at least one antiarrhythmic drug;
3. Prepared to undergo atrial fibrillation catheter ablation;
4. Provide informed consent to participate in the study, comply with follow-up trials and evaluation procedures.

Exclusion Criteria:

1. Presence of acute conditions such as acute phase after myocardial infarction (within 3 months), acute heart failure or new onset of cerebral infarction within 3 months;
2. On the heart transplant list;
3. Life expectancy less than 1 year;
4. With other bleeding disorders that cannot be treated with anticoagulation therapy;
5. With left atrial thrombus;
6. Heart failure with NYHA class III-IV or LVEF<40%;
7. With uncontrolled malignant tumor;
8. Obvious liver or kidney dysfunction (ALT, AST levels more than 2 times the upper limit of normal, and/or CCr<50%);
9. History of catheter radiofrequency ablation for atrial fibrillation or cardiac surgery;
10. Women who are pregnant, breastfeeding, planning to become pregnant, or of childbearing age but not using reliable contraception.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmias | 3 and 12 months from the date of procedure
  Efficacy endpoint:
  Including recurrence of atrial fibrillation, atrial flutter, and atrial tachycardia (sustaining more than 30s)

SECONDARY OUTCOMES:
Procedural complications | through study completion, an average of 1 year
  Safety endpoint:
  Occurrence of of atrioesophageal fistula, pulmonary vein stenosis, pericardial tamponade, phrenic nerve injury, and embolism

CONTACTS AND LOCATIONS:
Overall Officials: Yigang LI, Dr., Principal Investigator — Xinhua Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen M, Li C, Liao P, Cui X, Tian W, Wang Q, Sun J, Yang M, Luo L, Wu H, Li YG. Epidemiology, management, and outcomes of atrial fibrillation among 30 million citizens in Shanghai, China from 2015 to 2020: A medical insurance database study. Lancet Reg Health West Pac. 2022 May 3;23:100470. doi: 10.1016/j.lanwpc.2022.100470. eCollection 2022 Jun. PMID 35542895
- [Result] Hylek EM, Go AS, Chang Y, Jensvold NG, Henault LE, Selby JV, Singer DE. Effect of intensity of oral anticoagulation on stroke severity and mortality in atrial fibrillation. N Engl J Med. 2003 Sep 11;349(11):1019-26. doi: 10.1056/NEJMoa022913. PMID 12968085
- [Result] Sun J, Chen M, Wang Q, Zhang PP, Li W, Zhang R, Mo BF, Han B, Li XJ, Du W, Zhao L, Wang H, Yang B, Wu Y, Cai X, Li C, Chen TZ, Li YG. Adding six short lines on pulmonary vein isolation circumferences reduces recurrence of paroxysmal atrial fibrillation: Results from a multicenter, single-blind, randomized trial. Heart Rhythm. 2022 Mar;19(3):344-351. doi: 10.1016/j.hrthm.2021.11.014. Epub 2021 Nov 12. PMID 34775069
- [Result] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Result] Clarke JD, Piccini JP, Friedman DJ. The role of posterior wall isolation in catheter ablation of persistent atrial fibrillation. J Cardiovasc Electrophysiol. 2021 Sep;32(9):2567-2576. doi: 10.1111/jce.15164. Epub 2021 Jul 21. PMID 34258794
- [Result] Sugumar H, Thomas SP, Prabhu S, Voskoboinik A, Kistler PM. How to perform posterior wall isolation in catheter ablation for atrial fibrillation. J Cardiovasc Electrophysiol. 2018 Feb;29(2):345-352. doi: 10.1111/jce.13397. Epub 2017 Dec 26. PMID 29178497
- [Result] Cutler MJ, Johnson J, Abozguia K, Rowan S, Lewis W, Costantini O, Natale A, Ziv O. Impact of Voltage Mapping to Guide Whether to Perform Ablation of the Posterior Wall in Patients With Persistent Atrial Fibrillation. J Cardiovasc Electrophysiol. 2016 Jan;27(1):13-21. doi: 10.1111/jce.12830. Epub 2015 Oct 30. PMID 26515166
- [Result] Bai R, Di Biase L, Mohanty P, Trivedi C, Dello Russo A, Themistoclakis S, Casella M, Santarelli P, Fassini G, Santangeli P, Mohanty S, Rossillo A, Pelargonio G, Horton R, Sanchez J, Gallinghouse J, Burkhardt JD, Ma CS, Tondo C, Natale A. Proven isolation of the pulmonary vein antrum with or without left atrial posterior wall isolation in patients with persistent atrial fibrillation. Heart Rhythm. 2016 Jan;13(1):132-40. doi: 10.1016/j.hrthm.2015.08.019. Epub 2015 Aug 13. PMID 26277862
- [Result] O'Neill L, Hensey M, Nolan W, Keane D. Clinical outcome when left atrial posterior wall box isolation is included as a catheter ablation strategy in patients with persistent atrial fibrillation. J Interv Card Electrophysiol. 2015 Oct;44(1):63-70. doi: 10.1007/s10840-015-0024-2. Epub 2015 Jun 12. PMID 26066661
- [Result] Liu X, Gao X, Chen L, Shen L, Liu M, Xu Y. Clinical impact of posterior wall isolation in catheter ablation for persistent atrial fibrillation: A systematic review and meta-analysis. Pacing Clin Electrophysiol. 2022 Oct;45(10):1268-1276. doi: 10.1111/pace.14591. Epub 2022 Sep 20. PMID 36073753
- [Result] Lee JM, Shim J, Park J, Yu HT, Kim TH, Park JK, Uhm JS, Kim JB, Joung B, Lee MH, Kim YH, Pak HN; POBI-AF Investigators. The Electrical Isolation of the Left Atrial Posterior Wall in Catheter Ablation of Persistent Atrial Fibrillation. JACC Clin Electrophysiol. 2019 Nov;5(11):1253-1261. doi: 10.1016/j.jacep.2019.08.021. Epub 2019 Oct 30. PMID 31753429
- [Result] Kistler PM, Chieng D, Sugumar H, Ling LH, Segan L, Azzopardi S, Al-Kaisey A, Parameswaran R, Anderson RD, Hawson J, Prabhu S, Voskoboinik A, Wong G, Morton JB, Pathik B, McLellan AJ, Lee G, Wong M, Finch S, Pathak RK, Raja DC, Sterns L, Ginks M, Reid CM, Sanders P, Kalman JM. Effect of Catheter Ablation Using Pulmonary Vein Isolation With vs Without Posterior Left Atrial Wall Isolation on Atrial Arrhythmia Recurrence in Patients With Persistent Atrial Fibrillation: The CAPLA Randomized Clinical Trial. JAMA. 2023 Jan 10;329(2):127-135. doi: 10.1001/jama.2022.23722. PMID 36625809
- [Result] Pambrun T, Duchateau J, Delgove A, Denis A, Constantin M, Ramirez FD, Chauvel R, Tixier R, Welte N, Andre C, Nakashima T, Nakatani Y, Kamakura T, Takagi T, Krisai P, Cheniti G, Vlachos K, Bourier F, Takigawa M, Kitamura T, Frontera A, Sacher F, Hocini M, Jais P, Haissaguerre M, Walton RD, Derval N. Epicardial course of the septopulmonary bundle: Anatomical considerations and clinical implications for roof line completion. Heart Rhythm. 2021 Mar;18(3):349-357. doi: 10.1016/j.hrthm.2020.11.008. Epub 2020 Nov 11. PMID 33188900
- [Result] Thiyagarajah A, Kadhim K, Lau DH, Emami M, Linz D, Khokhar K, Munawar DA, Mishima R, Malik V, O'Shea C, Mahajan R, Sanders P. Feasibility, Safety, and Efficacy of Posterior Wall Isolation During Atrial Fibrillation Ablation: A Systematic Review and Meta-Analysis. Circ Arrhythm Electrophysiol. 2019 Aug;12(8):e007005. doi: 10.1161/CIRCEP.118.007005. Epub 2019 Aug 12. PMID 31401853
- [Result] Valderrabano M, Peterson LE, Swarup V, Schurmann PA, Makkar A, Doshi RN, DeLurgio D, Athill CA, Ellenbogen KA, Natale A, Koneru J, Dave AS, Giorgberidze I, Afshar H, Guthrie ML, Bunge R, Morillo CA, Kleiman NS. Effect of Catheter Ablation With Vein of Marshall Ethanol Infusion vs Catheter Ablation Alone on Persistent Atrial Fibrillation: The VENUS Randomized Clinical Trial. JAMA. 2020 Oct 27;324(16):1620-1628. doi: 10.1001/jama.2020.16195. PMID 33107945
- [Result] He Z, Yang L, Bai M, Yao Y, Zhang Z. Feasibility, efficacy, and safety of ethanol infusion into the vein of Marshall for atrial fibrillation: A meta-analysis. Pacing Clin Electrophysiol. 2021 Jul;44(7):1151-1162. doi: 10.1111/pace.14263. Epub 2021 May 24. PMID 33990979
- [Result] Chen M, Sun J, Wang QS, Zhang PP, Li W, Zhang R, Mo BF, Yu YC, Cai X, Yang M, Lian XM, Zhao Y, Gong C, Yu Y, Liu B, Feng X, Lu Q, Li YG. Long-term outcome of combined catheter ablation and left atrial appendage closure in atrial fibrillation patients. Int J Cardiol. 2022 Dec 1;368:41-48. doi: 10.1016/j.ijcard.2022.08.007. Epub 2022 Aug 8. PMID 35952939
- [Result] Mo BF, Sun J, Zhang PP, Li W, Chen M, Yuan JL, Yu Y, Wang QS, Li YG. Combined Therapy of Catheter Ablation and Left Atrial Appendage Closure for Patients with Atrial Fibrillation: A Case-Control Study. J Interv Cardiol. 2020 Jun 25;2020:8615410. doi: 10.1155/2020/8615410. eCollection 2020. PMID 32669982
- [Result] Lin H, Chen YH, Hou JW, Lu ZY, Xiang Y, Li YG. Role of contact force-guided radiofrequency catheter ablation for treatment of atrial fibrillation: A systematic review and meta-analysis. J Cardiovasc Electrophysiol. 2017 Sep;28(9):994-1005. doi: 10.1111/jce.13264. Epub 2017 Jun 23. PMID 28569422